CLINICAL TRIAL: NCT05786443
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Safety, Tolerability, and Preliminary Efficacy of Empagliflozin Among Patients Initiating Hemodialysis for the Treatment of End-Stage Kidney Disease
Brief Title: Safety and Efficacy of Empagliflozin in Hemodialysis
Acronym: SEED
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22-01497
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental): Participants with end-stage kidney disease (ESRD) initiating hemodialysis will receive Empagliflozin 10 mg daily for 12 weeks.
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator): Participants with ESRD initiating hemodialysis will receive Empagliflozin-matching placebo daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Sodium glucose cotransporter 2 inhibitor (SGLT2i) dosed once-daily over 12 weeks. Administered as oral tablet.
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo — Empagliflozin-matching placebo dosed once-daily over 12 weeks. Administered as oral tablet.
  Arms: Placebo

SUMMARY:
A 12-week, phase II, randomized, double-blind, placebo-controlled, multi-center study to assess the safety, tolerability, and preliminary efficacy of empagliflozin versus placebo among patients initiating hemodialysis (n=60) for the treatment of end-stage kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years on maintenance hemodialysis (HD) with residual kidney function
* Thrice-weekly HD
* Willingness and capacity to provide informed consent
* For women of childbearing potential, a negative pregnancy test is required at screening

Exclusion Criteria:

* Does not have capacity to consent
* Anuria (daily urine volume < 200 mL/day)
* Planned kidney transplant within 3 months
* Recurrent urinary tract infections (>2 episodes/year or antibiotic prophylaxis)
* New York Heart Association (NYHA) Class IV heart failure (HF)
* Myocardial infarction, unstable angina, revascularization procedure (e.g., stent or bypass graft surgery), or cerebrovascular accident within 12 weeks
* History of diabetic ketoacidosis
* Type 1 Diabetes Mellitus
* Hereditary glucose-galactose malabsorption or primary renal glucosuria
* Liver disease (e.g., acute hepatitis, chronic active hepatitis, cirrhosis); Alanine aminotransferase (ALT) levels >2.0 times the upper limit of normal (ULN) or total bilirubin >1.5 times the ULN, unless consistent with Gilbert's disease
* Active malignancy (exceptions: squamous and basal cell carcinomas of the skin and carcinoma of the cervix in situ) defined as malignancy under active treatment with chemotherapy, radiation or immunotherapy, or being treated as palliative.
* Major surgery within 12 weeks
* Atraumatic amputation within past 12 months of screening, or an active skin ulcer, osteomyelitis, gangrene, or critical ischemia of the lower extremity within 6 months of screening
* Combination use of angiotensin-converting enzyme inhibitor (ACEi) and angiotensin receptor blocker (ARB)
* Current use of an SGLT2 inhibitor (within 6 weeks prior to randomization)
* Known allergies, hypersensitivity, or intolerance to SGLT2i or its excipients
* Received an active investigational drug (including vaccines) other than a placebo agent, or used an investigational medical device within 12 weeks before Day 1/baseline
* Pregnant or breast-feeding or planning to become pregnant or breast-feed during the study
* Women of childbearing potential not willing to use a highly-effective method(s) of birth control, or who are unwilling or unable to be tested for pregnancy.
* Any condition that in the opinion of the investigator would make participation not in the best interest of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Extracellular Volume from Baseline to 12 Weeks | Baseline, Week 12
  Extracellular volume is the sum of the plasma volume and interstitial fluid volume.
Change in Intracellular Volume from Baseline to 12 Weeks | Baseline, Week 12
  Intracellular volume is the fluid content within the body's cells.
Change in Total Body Water from Baseline to 12 Weeks | Baseline, Week 12
Change in 24-Hour Urine Volume from Baseline to 12 Weeks | Baseline, Week 12
  Urine volume over a 24-hour period.

SECONDARY OUTCOMES:
Change in 24-Hour Urine Albumin Excretion from Baseline to 12 Weeks | Baseline, Week 12
  Albumin excreted in the urine over a 24-hour period.
Change in 24-Hour Ambulatory Blood Pressure from Baseline to 12 Weeks | Baseline, Week 12
  Blood pressure measured over a 24-hour period.
Change in Heart Rate Variability from Baseline to 12 Weeks | Baseline, Week 12
  Variance in time between the heart beats.
Incidence of Intra-Dialytic Hypotension | Up to Week 12
  Intra-dialytic hypotension defined as nadir systolic blood pressure (SBP) <90 mmHg if pre-HD SBP≤160 mmHg, or nadir SBP <100 mmHg if pre-HD SBP >160 mmHg.
Incidence of Inter-Dialytic Hypotension | Up to Week 12
  Inter-dialytic hypotension defined symptomatic SBP <90 mmHg or hypotension requiring adjustment in blood pressure medications or treatment in an emergency or hospitalized setting.
Incidence of Serious Hypotension | Up to Week 12
  Defined as hypotension requiring hospitalization, emergency room (ER) visit, or reduction of blinded study medication or other anti-hypertensive medications.
Incidence of Non-Serious Hypoglycemia | Up to Week 12
  Detected via clinical lab data.
Incidence of Serious Hypoglycemia | Up to Week 12
  Defined as hypoglycemia requiring hospitalization, emergency room (ER) visit or the combination of glucose<70 mg/dL and urgent glucagon or carbohydrate use.
Incidence of Ketoacidosis | Up to Week 12
  Defined as metabolic state associated with pathologically high serum and urine concentrations of ketone bodies.
Number of Adverse Events | Up to Week 12
Number of Serious Adverse Events | Up to Week 12

OTHER OUTCOMES:
Recruitment Rate | Up to Week 12
  Defined as average number of patients recruited per month.
Withdrawal Rate | Up to Week 12
  Defined as percentage of participants who withdraw before completing the trial.
Percentage of Participants Lost to Follow-Up | Up to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: David Charytan, MS, MSc, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: David.Charytan@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to David.Charytan@nyulangone.org . To gain access, data requestors will need to sign a data access agreement.